CLINICAL TRIAL: NCT03315962
Title: Simplified Isoniazid Preventive Therapy (SPIRIT) Strategy to Reduce TB Burden
Brief Title: Simplified Isoniazid Preventive Therapy Strategy to Reduce TB Burden
Acronym: SEARCH-IPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Makerere University (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Cipla Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-21030; R01AI125000 (NIH)
Record Dates: First submitted 2017-09-26; First posted 2017-10-20 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis; HIV/AIDS
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 1: DHO Intervention Arm (Experimental): A selection of DHO or TB district supervisors that are randomized to the multicomponent SPIRIT intervention.
  Interventions: Behavioral: SPIRIT Intervention
- Aim 1: DHO Control Arm (No Intervention): A selection of DHO or TB district supervisors that are randomized to the country standard of care, but not to receive the study intervention.

INTERVENTIONS:
Behavioral: SPIRIT Intervention — The intervention will include implementing a teaching collaborative among group of DHOs and TB Supervisors, enabling text messaging between DHOs and front line providers, and establishing a report collaborative where DHOs will receive feedback on the performance of their district in administering IPT compared to other districts.
  Arms: Aim 1: DHO Intervention Arm

SUMMARY:
The overall objective of this study is to determine if a multi-component implementation intervention (SPIRIT) and additional leadership and management training that targets District Health Officers (DHOs) can increase IPT initiation among HIV-infected persons, as compared to country standard practices, in a cluster randomized trial in Uganda.

DETAILED DESCRIPTION:
The failure to use isoniazid (INH) preventative therapy (IPT) in HIV-infected individuals in Sub-Saharan Africa represents one of the single biggest implementation gaps between evidence and practice in today's response to the HIV epidemic. The proposed study will evaluate the effectiveness of a multi-component intervention to improve IPT uptake in two regions of Uganda. The study design is a randomized controlled trial (RCT) where the unit of randomization is clusters of districts in Uganda. The clusters consist of 5-7 districts and the District Health Officer (DHO) and District TB and Leprosy Supervisor (DTLS) from each district is invited to participate. The SPIRIT intervention is based on the PRECEDE framework which outlines the importance of social networks, social influence, and behavior change.

The SEARCH-IPT multi-component intervention includes:

* A teaching collaborative which will be formed within the randomized clusters of district DHOs and DTLSs to create a mini-collaborative, which will be led by an opinion leader with HIV and TB expertise, to spread new scientific knowledge about IPT and the clinical ability to rule out TB, and to facilitate discussion between DHOs.
* A "toolkit" of options to ease IPT implementation will support DHOs to scale up IPT through the study of the comparative effectiveness of material contributions to their day-to-day function of managing front line providers and clinics.
* A reporting collaborative comprised of the teaching collaborative groups, will define targets as a group, and reconvening every 6 months for 3 years (with the additional option of 36 months for a final report back), where each collaborative has an opportunity to share progress and results.

In addition, an enhanced business training & 'training-of-trainers' curriculum will be conducted to evaluate the effect of enhanced business training among intervention group DHOs from Phase 1 (Years 1-3 of trial follow-up) in the southwestern Uganda region on IPT initiation during years 4-5 of trial follow-up (Phase 2).

ELIGIBILITY:
AIM 1 - Spirit Intervention:

Inclusion Criteria:

* District Health Officer or TB District Supervisor (or other DHO-appointed TB focal person) in Uganda.
* By definition, the DHO or TB District Supervisor are all ≥18 years of age.

Exclusion Criteria:

* Planned departure from position as DHO or TB District Supervisor prior to randomization.
* DHOs from Kampala and Wakiso districts, Uganda.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Havlir, MD, Principal Investigator — University of California, San Francisco; Gabriel Chamie, MD, MPH, Study Chair — University of California, San Francisco
Locations (1):
- Infectious Diseases Research Collaboration, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kakande E, Christian C, Balzer LB, Owaraganise A, Nugent JR, DiIeso W, Rast D, Kabami J, Johnson Peretz J, Camlin CS, Shade SB, Geng EH, Kwarisiima D, Kamya MR, Havlir DV, Chamie G. A mid-level health manager intervention to promote uptake of isoniazid preventive therapy among people with HIV in Uganda: a cluster randomised trial. Lancet HIV. 2022 Sep;9(9):e607-e616. doi: 10.1016/S2352-3018(22)00166-7. Epub 2022 Jul 28. PMID 35908553
- [Derived] Johnson-Peretz J, Christian C, Akatukwasa C, Atwine F, Kamya MR, Havlir DV, Chamie G, Camlin CS, Kakande E. Small-world challenges and solutions identified by mid-level managers within a decentralised healthcare system during a qualitative sub-study of a tuberculosis-prevention therapy rollout intervention in Uganda: "When a big drum like the District Health Officer talks". Res Sq [Preprint]. 2025 Jul 31:rs.3.rs-5046392. doi: 10.21203/rs.3.rs-5046392/v1. PMID 40766233
- [Derived] Christian C, Kakande E, Nahurira V, Akatukwasa C, Atwine F, Bakanoma R, Itiakorit H, Owaraganise A, DiIeso W, Rast D, Kabami J, Peretz JJ, Shade SB, Kamya MR, Havlir DV, Chamie G, Camlin CS. Mid-level managers' perspectives on implementing isoniazid preventive therapy for people living with HIV in Ugandan health districts: a qualitative study. BMC Health Serv Res. 2024 Mar 8;24(1):313. doi: 10.1186/s12913-024-10803-9. PMID 38454501

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: clusters of DHOs
Period: Overall Study
Arm/Group | Aim 1: DHO Intervention Arm | Aim 1: DHO Control Arm
Started | 86; 7 clusters of DHOs | 77; 7 clusters of DHOs
Completed | 86; 7 clusters of DHOs | 77; 7 clusters of DHOs
Not Completed | 0; 0 clusters of DHOs | 0; 0 clusters of DHOs

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aim 1: DHO Intervention Arm | Aim 1: DHO Control Arm | Total
Number analyzed (Participants) | 86 | 77 | 163
Age, Customized [Count of Participants; unit: Participants] — Population: Age at Baseline was not collected
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 78 | 71 | 149
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 86 | 77 | 163
Region of Enrollment [Number; unit: participants]
  Uganda | 86 | 77 | 163

OUTCOME MEASURES:

1. Primary Outcome: IPT Initiation Rate
Description: Incident rate of IPT initiation (events per person-year) among adults with HIV in facilities overseen by participants. Mean was calculated as the average rate across the clusters (groups of DHOs)
Time Frame: 2 years
Population: Adults with HIV in facilities overseen by DHOs in 14 clusters (between 4 and 7 districts per cluster), based on geographical adjacency, number of urban versus rural districts, number of people with HIV in care, and region. Clusters were pair-matched on characteristics expected to be predictive of IPT initiation: region, number of adults in HIV care, presence of large urban centres, and a community that had participated from 2013 to 2017 in the SEARCH HIV test-and-treat trial (NCT01864603).
Measure: Mean (95% Confidence Interval); unit: events per person-years
Units Other Than Participants: clusters of DHOs
Arm/Group | Aim 1: DHO Intervention Arm | Aim 1: DHO Control Arm
Number analyzed (Participants) | 86 | 77
Number analyzed (clusters of DHOs) | 7 | 7
events per person-years | 0.74 [0.59 to 0.88] | 0.65 [0.55 to 0.75]

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Aim 1: DHO Intervention Arm | Aim 1: DHO Control Arm
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/77
Other Adverse Events (participants affected / at risk) | 0/86 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/62/NCT03315962/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT03315962/SAP_001.pdf